CLINICAL TRIAL: NCT02407847
Title: The (Cost-)Effectiveness of Substitution in Out-of-hours Primary Care; Towards an Optimal Balance Between General Practitioners and Nurse Practitioners.
Brief Title: The Effect of Substitution of Out-of-hours Care From General Practitioners to Nurse Practitioners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Stichting Kwaliteit en Ontwikkeling Huisartsenzorg (Other); Centrale Huisartsenpost Eindhoven (CHP) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VS_in_spoedzorg
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Out-of-hours Care Services; Primary Healthcare
Keywords: Nurse practitioners; Primary healthcare; Emergency Medical Services; Substitution of care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Practitioners Care (No Intervention): Usual medical care provided by General Practitioners at the Primary Out-of-Hours Service.
- Nurse Practitioners Care (Experimental): Medical care provided by both Nurse Practitioners and General Practitioners at the Primary Out-of-Hours Service.
  Interventions: Other: care provided by Nurse Practitioners

INTERVENTIONS:
Other: care provided by Nurse Practitioners — Patients will receive care at the Primary Out of Hours Emergency Service by a Nurse Practitioner instead of a General Practitioner (substitution of care from physicians to nurses).
  Arms: Nurse Practitioners Care

SUMMARY:
The aim of this study is to explore the effects of substitution in out-of-hours primary care. In consecutive stages an extra General Practitioner (GP) is substituted by a Nurse Practitioner (NP) aiming at replacing 3 out of 4 GPs by NPs. Effects are measured in terms of feasibility and cost-efficiency.

DETAILED DESCRIPTION:
Out-of-hours care in the Netherlands is under pressure. Workload for GPs during out-of-hours care is high and there are concerns about maintaining the quality of care. Since 80% of the complaints shown in out-of-hours care is neither complex nor urgent not all patients necessarily have to be seen by a GP.

A previous study (ID: 80-82800-98-227) indicated that shifting care from GPs to NPs is possible in terms of safety and quality of care and resulted in cost savings due to less treatment. In that study 4 GPs and 1 NP provided care in the experimental condition and 5 GPs provided care in the control condition. Based on the results it is hypothesized that NPs are competent to diagnose and treat at least 75% of the complaints shown in out-of-hours primary care. Substituting more GPs by NPs in out-of-hours care will probably lead to more cost savings.

In the current study care delivered and direct healthcare costs are compared between different team compositions. In the experimental condition care is provided by a team of NPs and GPs. The intervention starts with a team of 4 professionals in both the experimental (3 GPs and 1 NP) and the control (4 GPs) condition; in consecutive stages an extra GP is substituted by an NP aiming at replacing 3 out of 4 GPs with by NPs.

Control: 4 GPs

Stage 1: experimental: 3 GPs & 1 NP

Stage 2: experimental: 2 GPs & 2 NPs

Stage 3: experimental: 1 GP & 3 NPs

Both feasibility and cost-efficiency will lead to recommendations on the optimal balance in a team between GPs and NPs.

ELIGIBILITY:
Inclusion Criteria:

* Patients (with urgencylevel U2, U3, U4, or U5) requesting an appointment at the primary out-of-hours service during the weekend between 10am and 6pm.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9647 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The number of consultations per healthcare provider. | 18 months
  To measure substitution of healthcare, the number of consultations per in the experimental and control group, and per healthcare provider will be measured. These data will be derived from electronic medical records.

SECONDARY OUTCOMES:
Number and characteristics of patients and experienced workload. | 18 months
  Objective workload will be measured by the numbers of consults, taking into account the urgency levels of the complaints and type of complaint. These data will be derived from electronic medical records. Subjective workload will be measured by interviews and focusgroups.
Direct healthcare costs related to care provide by NPs and GPs will be calculated. | 18 months
  Costs related to care provided in the experimental and control group, and per discipline will be calculated, including number of consultations, resource use, referrals, and prescriptions.
Patient characteristics (composite) | 18 months
  Patient characteristics of patients seen in the experimental and control group and per healthcare provider include age, gender, urgency and type of complaint. These data will be derived from electronic medical records.
The number of prescriptions; number of test & investigations ordered and referral to the emergency department. | 18 months
  The performance of the two conditions as well as the healthcare providers will be measures by number of prescriptions; number of test & investigations ordered and referral to the emergency department. These data will be derived from electronic medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Centrale Huisartsen Post (CHP), Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Derived] van der Biezen M, Wensing M, van der Burgt R, Laurant M. Towards an optimal composition of general practitioners and nurse practitioners in out-of-hours primary care teams: a quasi-experimental study. BMJ Open. 2017 May 30;7(5):e015509. doi: 10.1136/bmjopen-2016-015509. PMID 28559458